CLINICAL TRIAL: NCT03427840
Title: Efficacy of Intraoperative Superior Hypogastric Plexus Blockade for Postoperative Pain in Laparoscopic Hysterectomy
Brief Title: Superior Hypogastric Plexus Blockade in Laparoscopic Hysterectomy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Derince Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Hande G. Aytuluk, M.D., Principal investigator, Derince Training and Research Hospital
Other Study IDs: U1111-1208-8608
Record Dates: First submitted 2018-02-01; First posted 2018-02-09 (Actual); Last update posted 2018-03-20 (Actual); Status verified 2018-03

CONDITIONS: Superior Hypogastric Plexus Block; Hysterectomy; Minimally Invasive Surgery; Laparoscopy; Pain, Postoperative; Gynecologic Disease
Keywords: Superior Hypogastric Plexus Block; Hysterectomy; Minimally invasive surgery; Laparoscopy; Pain; Gynecologic Disease
MeSH Terms: conditions — Pain, Postoperative; Genital Diseases, Female; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hypo: The participants with a superior hypogastric block
  Interventions: Procedure: Procedure/Surgery: superior hypogastric block
- NoHypo: The participants without a superior hypogastric block; the patients with an epidural catheter, who receive a different block technique (ie: TAP block), or who are unsuitable for SHP block (ie: if retroperitone is opened intraoperatively by the surgeon)

INTERVENTIONS:
Procedure: Procedure/Surgery: superior hypogastric block — superior hypogastric blockade during surgery
  Groups: Hypo

SUMMARY:
The primary indication for superior hypogastric plexus (SHP) block is visceral pelvic pain, most commonly from malignancy of the ovary, uterus, cervix, bladder, rectum or prostate. Per-cutaneous SHP blocks should be done under guidance of ultrasonography, fluoroscopy, magnetic resonance or computed tomography. During minimally invasive laparoscopic surgery, percutaneous technique can be done under the guidance of cameras.

DETAILED DESCRIPTION:
Laparoscopic surgeries have many advantages over open surgeries. Laparoscopic procedures are mostly preferred for surgical treatment of gynecologic diseases, because of best cosmetically results, less perioperative complications, early recovery, and less postoperative pain.

There are many undesirable effects of systemic reactions to the pain. Accordingly, multi-modal analgesic approach (including nerve blocks) for postoperative acute pain can decrease the side effects of the drugs (especially opioids) significantly.

The primary indication for superior hypogastric plexus (SHP) block is visceral pelvic pain, most commonly from malignancy of the ovary, uterus, cervix, bladder, rectum or prostate. Per-cutaneous SHP blocks should be done under guidance of ultrasonography, fluoroscopy, magnetic resonance or computed tomography. During minimally invasive laparoscopic surgery, per-cutaneous technique can be done under the guidance of cameras.

SHP block has been performed by anesthetists or surgeons in Kocaeli Derince Training and Research Hospital regularly since they have discovered the advantages of this block technique. SHP can be useful to decrease postoperative pain scores and opioid or NSAID consumption significantly.

ELIGIBILITY:
Inclusion Criteria:

* ASA I - II
* Elective laparoscopic hysterectomy

Exclusion Criteria:

* ASA III
* Different kind of surgery
* Known allergy to local anesthetic drugs
* Different analgesia protocol (ie: epidural, TAP block,..)
* Refusal of the patient

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — patients who are scheduled for hysterectomy
Study Population: The patients who are scheduled for elective laparoscopic hysterectomy under general anesthesia.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2018-03-18 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-07-01 (Estimated)

PRIMARY OUTCOMES:
postoperative pain scores (PACU) | 1 hour (postoperatively)
  Patients' pain scores will be scored with a 10 cm Visual Analogue Scale (VAS). Each will be scored between 0-10 (0: no pain; 10: worst pain ever)
postoperative opioid/NSAID consumption (PACU) | 1 hour (postoperatively)
  nonsteroid antiinflammatory drugs (NSAID) or opioid drugs that are applied to patients will be noted down.
rescue analgesic time | 48 hours (first analgesic demand time will be noted down)
  Time to first analgesic demand at gynecology ward (after transfer from PACU to gynecology ward)
postoperative pain scores (ward) | 48 hours (postoperatively)
  Patients' pain scores will be scored with a 10 cm Visual Analogue Scale (VAS). Each will be scored between 0-10 (0: no pain; 10: worst pain ever)
postoperative opioid/NSAID consumption (ward) | 48 hours (total)
  NSAID or opioid drugs that are applied to patients will be noted down. Target VAS score for NSAID is >4; if there is no response to NSAID and pain is worsening opioid drugs will be applied

SECONDARY OUTCOMES:
Intraoperative hemodynamics | from SHP block to the end of the surgery (approximately 15 min)
  (If the patient is received a SHP block intraoperatively) post-block hemodynamical parametres will be noted down
length of stay | 3-5 days (expected)
  length of hospital stay time will be noted
complications due to SHP block | 3-5 days (from surgery to discharge from the hospital)
  intra/postoperative complications will be noted. (ie: intra-vascular local anesthetic injection, vascular puncture, hemodynamical changes after injection,.. )

CONTACTS AND LOCATIONS:
Overall Officials: Hande Aytuluk, MD, Principal Investigator — Derince Training and Research Hospital; Ahmet Kale, Prof, Study Chair — Derince Training and Research Hospital; Gulfem Basol, MD, Study Chair — Derince Training and Research Hospital
Locations (1):
- Derince Training and Research Hospital, Kocaeli, Derince, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The investigators do not prefer to share the study plan and records.

REFERENCES:
- [Result] Song T, Kim MK, Jung YW, Yun BS, Seong SJ, Choi CH, Kim TJ, Lee JW, Bae DS, Kim BG. Minimally invasive compared with open surgery in patients with borderline ovarian tumors. Gynecol Oncol. 2017 Jun;145(3):508-512. doi: 10.1016/j.ygyno.2017.03.019. Epub 2017 Apr 2. PMID 28381342
- [Result] Lovich-Sapola J, Smith CE, Brandt CP. Postoperative pain control. Surg Clin North Am. 2015 Apr;95(2):301-18. doi: 10.1016/j.suc.2014.10.002. Epub 2015 Jan 24. PMID 25814108
- [Result] Sindt JE, Brogan SE. Interventional Treatments of Cancer Pain. Anesthesiol Clin. 2016 Jun;34(2):317-39. doi: 10.1016/j.anclin.2016.01.004. PMID 27208713
- [Result] Erdine S, Yucel A, Celik M, Talu GK. Transdiscal approach for hypogastric plexus block. Reg Anesth Pain Med. 2003 Jul-Aug;28(4):304-8. doi: 10.1016/s1098-7339(03)00191-3. PMID 12945023
- [Derived] Aytuluk HG, Kale A, Basol G. Laparoscopic Superior Hypogastric Blocks for Postoperative Pain Management in Hysterectomies: A New Technique for Superior Hypogastric Blocks. J Minim Invasive Gynecol. 2019 May-Jun;26(4):740-747. doi: 10.1016/j.jmig.2018.08.008. Epub 2018 Aug 28. PMID 30165185